CLINICAL TRIAL: NCT04757896
Title: Comparison of Ultrasound Guided Medial Approach and Lateral Approach of the Costoclavicular Blockage: A Prospective Randomised Study
Brief Title: Costoclavicular Blockage for Upper Limb Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ilker Ince, Assoc. Prof. Dr. İlker İNCE, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/540
Record Dates: First submitted 2021-02-01; First posted 2021-02-17 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Anesthesia
Keywords: brachial plexus block

STUDY DESIGN:
Intervention Model Description: Assignment
Masking Description: blind surgeon and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costoclavicular block lateral aproach (Active Comparator): An 80-100 mm needle will be directed from the lateral to the medial with the ultrasound guided in-plane technique and the blockage procedure will be completed by injecting
  Interventions: Procedure: Lateral costoclavicular approach
- Costoclavicular block medial aproach (Active Comparator): An 80-100 mm needle will be directed from the medial to the lateral with the ultrasound guided in-plane technique and the blockage procedure will be completed by injecting
  Interventions: Procedure: Medial costoclavicular approach

INTERVENTIONS:
Procedure: Lateral costoclavicular approach — USG guided lateral costoclavicular approach for brachial plexus block
  Arms: Costoclavicular block lateral aproach
Procedure: Medial costoclavicular approach — USG guided medial costoclavicular approach for brachial plexus block
  Arms: Costoclavicular block medial aproach

SUMMARY:
To evaluate the success of surgical anesthesia of lateral and medial approaches of the costoclavicular block in patients undergoing upper extremity surgery.

DETAILED DESCRIPTION:
Introduction:Upper limb surgeries are used on various pathology cases including tendon injuries, carpal tunnel syndrome, tenosynovitis, fractures secondary to trauma, contractures and vascular injuries. In many of such operations local anaesthesia becomes insufficient, and general or regional anaesthesia is required for comfort of the patient and the surgeon. Today, widespread use of nerve stimulators and ultrasound, the availability of post-operative pain management options, applicability of regional anaesthesia where there is risk of complications with general anaesthesia and its applicability along with general anaesthesia for pain management has made regional anaesthesia an attractive solution.The costoclavicular cavity lies in the depth and back of the median of clavicular. It connects to subclavius and clavicular terminus of pectoralis major muscle at the anterior and to the anterior chest wall at the posterior. The cavity is cranially continuous with the supraclavicular fossa and caudally continuous with the medial infraclavicular fossa above the upper border of the pectoralis minor muscle. Unlike the lateral infraclavicular fossa, the cords lie in the costoclavicular cavity in a relatively superficial form in a bundled triangular arrangement. Anatomical layout of cords in the costoclavicular cavity makes this an attractive area for ultrasound imaging and infraclavicular brachial plexus blockage. After placing the linear ultrasound probe on the midclavicular line and even in parallel to the clavicular, the three cords are imaged along with the axillary artery, whereupon local anaesthetic injection can be made with in-plane technique, directing the needle from lateral to medial.

Medial approach to costoclavicular block defined by Nieuwveld involves placement of the linear ultrasound probe on the midclavicular line in parallel with the clavicular, as in the lateral approach, followed by imaging of the three cords alongside the axillary artery, whereupon the needle is directed from the medial to the lateral with the in-plane technique and applying local anaesthetic injection to the midpoint of three cords.

The sample size calculation is done based on the time for establishing total anaesthesia and anaesthesia lead time variables in reference to the study conducted by Prangmalee Leurcharusmee et al. Calculating for 16±5 for lateral approach and 21±7 for medial approach, it is calculated that each group should include 44 patients at 80% power and 95% reliability rate for a meaningful difference at 5 minutes, requiring a total of 88 patients.After obtaining approval of the local ethics board, 88 patients who are considered for emergency or elective superior extremity surgery, in ASA I-IV group, in 18 to 75 age group, who do not have any known serious illness and who consent to participate will be included in the study.

Material and Method:Patients in ASA IV group and above, patients taking anticoagulant/antiaggregate treatments, patients with nervous disorders, patients with infections or open wounds at the operation area and patients with allergies against any drug to be used in the study will be excluded from the study.

Patients participating in the study will be randomly divided into 2 separate groups. These groups will be referred to as the Group M (Medial approach group) and Group L (Lateral approach group).

Patients will be reviewed before being taken to operating room, they will be informed regarding the considered operation and their consent will be taken. Patients will be moved to regional anaesthesia room before the operation, where they will be equipped with fingertip oxygen saturation monitoring and 20-22 gauge intravenous channel. After confirming operation area sterilisation will be done with skin antiseptic, the operation area will be covered with sterilised cover and linear USG probe will be prepared in sterile conditions. All procedures will be implemented by an experienced anaesthesiologist. A blind researcher will review the patients and the surgical team will also be kept blind regarding the type of procedure.

In Group M, after the patient will be taken to the regional anaesthesia room and preparations will be made, the blockage procedure will be applied by an anaesthesiologist who is not blind. The patient will be brought to supine position, the arm subject to procedure will be taken to 90° abduction with the palm looking at the ceiling. The Linear USG probe will be positioned on the midclavicular line and the chronometer will be started to record the scanning procedure time as the time elapsed until imaging of the axillary artery alongside with the three cords. After achieving optimum imaging skin infiltration will be applied with 1% lidocaine and an 80-100 mm needle will be directed from the medial to the lateral with the in-plane technique and the blockage procedure will be completed by injecting a combination of 10 cc 2% lidocaine and 10 cc 0.5% bupivacaine in the exact midpoint of the three cords.

In Group L, again the patient will be taken to the regional anaesthesia room and preparations will be made, and the blockage procedure will be applied by an anaesthesiologist who is not blind. The patient will be brought to supine position, the arm subject to procedure will be taken to 90° abduction with the palm looking at the ceiling. The Linear USG probe will be positioned on the midclavicular line and the chronometer will be started to record the scanning procedure time as the time elapsed until imaging of the axillary artery alongside with the three cords. After achieving optimum imaging skin infiltration will be applied with 1% lidocaine and an 80-100 mm needle will be directed from the medial to the lateral with the in-plane technique and the blockage procedure will be completed by injecting a combination of 10 cc 2% lidocaine and 10 cc 0.5% bupivacaine in the exact midpoint of the three cords.

The total procedure time, the complications arising during procedure, the local anaesthetic toxicity, the paraesthesia arising during the procedure, the distance between the needle tip and the pleura and the number of needle passes will be recorded for each procedure. A blind researcher will evaluate sensory blockage by checking radial, musculocutaneous, medial and ulnar nerve dermatomes with ice using triple point scale (0= no blockage, patient completely feels the cold; 1= analgesia, the patient does not feel the cold but feels the touch; 2= anaesthesia, the patient does not feel the touch) once per 5 minutes for 30/45 minutes taking the moment of needle removal as the 0 point. Motor block will also be evaluated by triple point scale (0=no blockage; 1=paraesthesia established; 2=paralysis established) once per 5 minutes for 30 minutes. Motor blockage at musculocutaneous, radial, median and ulnar nerves will be evaluated by elbow flexion, thumb abduction, thumb opposition and thumb adduction, in this order. Sensory and motor blockage starting time points and total anaesthesia establishment time points will be recorded. At 20/30 minutes point convex (M mode) USG probe will be used to evaluate diaphragmatic paralysis. Once surgical anaesthesia is established the operation will be started, the patient will be monitored throughout the operation, additional analgesia-sedation needs, returns to general anaesthesia and total surgery times will be recorded. After surgical operation is completed, patient and surgeon satisfaction will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergency upper limb surgery
* Between 18 to 80 years old
* ASA I-IV

Exclusion Criteria:

* <18 years old/ >80 Years old
* >ASA IV
* Any serious illness
* Anticoagulant/antiaggregate treatments
* Any allergies to the drugs that used in study
* İnfections or open wounds at the operation area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
success in providing surgical anesthesia via triple point scale evaluation | 30 minutes
  The triple point scale (0= no blockage, patient completely feels the cold; 1= analgesia, the patient does not feel the cold but feels the touch; 2= anaesthesia, the patient does not feel the touch) once per 5 minutes for 30/45 minutes taking the moment of needle removal as the 0 point. Motor block will also be evaluated by triple point scale (0=no blockage; 1=paraesthesia established; 2=paralysis established) once per 5 minutes for 30 minutes.

SECONDARY OUTCOMES:
Initiation time of block | 30 minutes
  Sensory and motor block initiation time

CONTACTS AND LOCATIONS:
Overall Officials: ataturk unıversity, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

REFERENCES:
- [Background] Karmakar MK, Sala-Blanch X, Songthamwat B, Tsui BC. Benefits of the costoclavicular space for ultrasound-guided infraclavicular brachial plexus block: description of a costoclavicular approach. Reg Anesth Pain Med. 2015 May-Jun;40(3):287-8. doi: 10.1097/AAP.0000000000000232. No abstract available. PMID 25899958
- [Background] Nieuwveld D, Mojica V, Herrera AE, Pomes J, Prats A, Sala-Blanch X. Medial approach of ultrasound-guided costoclavicular plexus block and its effects on regional perfussion. Rev Esp Anestesiol Reanim. 2017 Apr;64(4):198-205. doi: 10.1016/j.redar.2016.09.010. Epub 2016 Dec 9. English, Spanish. PMID 27938934
- [Background] Leurcharusmee P, Elgueta MF, Tiyaprasertkul W, Sotthisopha T, Samerchua A, Gordon A, Aliste J, Finlayson RJ, Tran DQH. A randomized comparison between costoclavicular and paracoracoid ultrasound-guided infraclavicular block for upper limb surgery. Can J Anaesth. 2017 Jun;64(6):617-625. doi: 10.1007/s12630-017-0842-z. Epub 2017 Feb 15. PMID 28205117